CLINICAL TRIAL: NCT03104114
Title: Evaluating Adherence and Persistence in Patients Receiving Oral Oncolytic Therapy in a Safety Net Hospital's Pharmacist-driven Medication Management Program
Brief Title: Pharmacist-led Intervention on Adherence in Patients Undergoing Treatment With an Oral Oncology Medication
Acronym: BSPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-35671
Record Dates: First submitted 2017-03-23; First posted 2017-04-07 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Adherence, Medication
MeSH Terms: conditions — Medication Adherence | interventions — Historically Controlled Study

STUDY DESIGN:
Intervention Model Description: Pharmacist-led intervention group vs historical-control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Historical Control (Placebo Comparator): Pharmacy care was standard, high-touch model where an institutional specialty pharmacy contact patients via telephone. Standard adherence and counseling was offered over the phone to patients.
  Interventions: Behavioral: Historical control
- Pharmacist-intervention (Experimental): In-person counseling with a clinical pharmacist prior and during treatment with an oral oncology medication. Patients meet with a clinical pharmacist prior, at month 3 and month 6 during the study.
  Interventions: Behavioral: pharmacist-intervention

INTERVENTIONS:
Behavioral: pharmacist-intervention — A clinical pharmacist provides patients with motivational counseling regarding their cancer treatments. Patients will be asked to complete three different surveys throughout the study; surveys focus on social support systems and both provider- and pharmacist-patient relationships
  Arms: Pharmacist-intervention
Behavioral: Historical control — Patients that did not receive in-person motivational counseling support from a clinical pharmacist prior and during treatment
  Arms: Historical Control

SUMMARY:
Boston Medical Center provides care to cancer patients on oral cancer medications through the use of Boston Medical Center Specialty Pharmacy (BMC SP). The use of oral medications in cancer treatments is relatively new and unfortunately, very little is known about adherence in cancer patients. This study will evaluate the influence of a pharmacist-driven medication management program on adherence and persistence rates. Boston Medical Center's Specialty Pharmacy Adherence Program (B-SPAP), will utilize a high-touch counseling model involving clinical pharmacist that will focus on educating patients about their oral cancer treatments. The program will require face-to-face counseling with a pharmacist, through the use of a proven patient teaching tool, prior to initiating treatment with oral oncolytic treatments and, periodically thereafter, based on protocol. This study will help improve our understanding of the role of the pharmacist in cancer patients. In addition, the study will help identify independent factors that may contribute or impact adherence. The outcomes of this program will be compared to a historical control group of patients that have already received treatment for their cancer through the BMC Specialty Pharmacy.

DETAILED DESCRIPTION:
Boston Medical Center's Specialty Pharmacy Adherence Program (B-SPAP) will focus on improving adherence and persistence through the implementation of a high-touch program. In order to be eligible for the program, patients must be initiated on oral chemotherapy or targeted therapy with a life expectancy >6 months. All patients will be administered a Patient Activation Measure (PAM) 13 survey prior to consultation. Patients eligible for our program will receive a 30-60 minute pharmacist consultation prior to initiation of treatment. The pharmacy consultation includes, but is not limited to the dissemination of medical information utilizing a standardized counseling checklist, supplying of patient education materials, pharmacist-led interventions, and/or the use of other materials or devices that may improve patient adherence. All counseling checklists and monitoring will be standardized and approved by a multidisciplinary oncology team. At week 1, 2, and 4, patients will be contacted by the pharmacist for an assessment of treatment goals; monthly contacts will continue thereafter by either a specialty pharmacist or certified pharmacy technician. Scheduled follow up visits with the consulting pharmacist will be made at months 3, 6 and 12. Prior to the scheduled pharmacist consultation, patients will be administered the PAM 13 survey. Patients with a treatment gap >37 days will be referred to the consulting pharmacist for follow up. The consulting pharmacist will attempt to contact the patient via telephone for an assessment of adherence and adverse drug-related events. If patients experience a treatment gap >45, then the patient will be contacted and scheduled for a pharmacist consultation, additionally, the prescribing provider will be notified. All consultations and interventions will be documented in the hospital's electronic medical record system, EPIC®.

ELIGIBILITY:
Pharmacist-intervention group

Inclusion Criteria:

1. Treatment with 1 or more oral oncology agents. Oral oncology agent defined as medication taken mouth with the purpose to treat a patient's cancer
2. Treatment dispensed through the BMC Specialty Pharmacy
3. Age>18 years
4. Life expectancy >6 months
5. Patients must have ability to give written consent, or, must have a legally authorized representative

Exclusion Criteria:

1. Treatment indicated for neoadjuvant, adjuvant, peri-operative treatment
2. Concurrent radiation treatment
3. Patients that are unable to have oral oncology agents dispense through BMC Specialty Pharmacy

Historical Control:

1. 2 controls:1 intervention match
2. Matched to a patient in intervention group based on drug type

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Medication Possession Ratio | Month 0(time of first dispense) to month 12 or discontinuation of medication, whichever occurs first
  MPR >80%
Persistence rate | Month 0(time of first dispense) to month 12 or discontinuation of medication, whichever occurs first
  allowance of 45 day time gap

SECONDARY OUTCOMES:
Health-belief model | Month 0(time of first dispense) to month 12 or discontinuation of medication, whichever occurs first
  PAM-13 surveys
Provider-patient relationship | Month 0(time of first dispense) to month 12 or discontinuation of medication, whichever occurs first
  Trust-in-physician survey
Pharmacist-patient relationship | Month 0(time of first dispense) to month 12 or discontinuation of medication, whichever occurs first
  Pharmacist satisfaction survey

CONTACTS AND LOCATIONS:
Overall Officials: scott gould, PharmD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No